CLINICAL TRIAL: NCT05744986
Title: The Systemic Effects of Transcatheter Renal Artery Sympathetic Denervation Using a Second- Generation Radiofrequency Ablation Catheter: A Multicenter Observational Study.
Brief Title: Transcatheter Renal Artery Sympathetic Denervation Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Gormin Tan, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2022.273
Record Dates: First submitted 2023-02-02; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Hypertension, Renal
Keywords: Resistant hypertension (rHT); sympathetic nervous system (SNS); endovascular renal denervation (RDN)
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SYMPICITY Spyral RENAL DENERVATION (RDN) SYSTEMTM — The second generation SYMPLICITY RDN catheterTM has 4 times electrodes that are arranged in spirally in 90-degree intervals. Theoretically, the newer generation catheter can provide more efficient and extensive denervation in a shorter period of time16. Its efficacy was confirmed in SYMPLICITY HTN ON-MED and OFF-MED trial, which confirmed a consistent and durable BP reduction that lasted into 36 months with or without adjuvant anti-hypertensive drugs

SUMMARY:
Hypertension is a common health problem that affects millions of people in the world. Poorly controlled blood pressure (BP) leads to cardiovascular, cerebrovascular and renal complications. Despite the availability of multitudes of anti-hypertensive drugs, the percentage of patients achieving optimal control of hypertension has remained disappointingly low.

Resistant hypertension (rHT) is defined as the failure to achieve target BP despite concurrent use of antihypertensive drugs of different classes, with one of them being diuretics. The reported prevalence of this condition ranged from 5 to 30%. Lifestyle modification, enhancing drug compliance, treating of secondary causes, or adding mineralocorticoid receptor antagonist such as spironolactone or eplerenone are well established strategies to treat resistant hypertension.

Besides factors such as, activated sympathetic nervous system (SNS) and increased sympathetic outflow was thought to contribute to the development of rHT as well. Autonomic sympathectomy by way of endovascular renal denervation (RDN) was once a hopeful candidate as an adjuvant treatment for patients with rHT and it had shown signals of efficacy in early trials. However, the blood-pressure lowering efficacy was not demonstrated in the larger-scaled, randomized, sham- controlled SYMPLICITY HTN-3 trial. One possible explanation of the lack of efficacy of RDN in this trial was the lower-than-expected BP responses in the RDN group and higher than-expected BP reduction in the control group which raised the speculation that some of the patients recruited were not true rHT as the trial intended to include. The suboptimal anti-hypertensive efficacy of RDN in HTN-3 was also partly attributed to the design of the first-generation RDN catheter, in which only a single electrode is deployed and might not offer sufficient sympathetic denervation as less than half of patients in the SYMPLICITY HTN-3 received 4 quadrants ablation.

The second generation SYMPLICITY RDN catheterTM has 4 times electrodes that are arranged in spirally in 90-degree intervals. Theoretically, the newer generation catheter can provide more efficient and extensive denervation in a shorter period of time. Its efficacy was confirmed in SYMPLICITY HTN ON-MED and OFF-MED trial, which confirmed a consistent and durable BP reduction that lasted into 36 months with or without adjuvant anti-hypertensive drugs.

BP reduction is only one of the effects of RDN. Previous observational studies of the first generation RDN catheter have shown an inconsistent effect of RDN in left ventricular (LV) remodelling, arrythmia modulation, arterial de-stiffening and quality of life. No report of these effects has been published with the newer generation catheter. Furthermore, vigorous efforts have been put into searching for clinical predictors that can identify patients in whom the BP reduction effect of RDN is most significant.

This study aims to investigate the systemic effects of RDN using the new generation SYMLICITY RDN catheterTM in patients with rHT.

DETAILED DESCRIPTION:
Hypertension is a common health problem that affects millions of people in the world. Poorly controlled blood pressure (BP) leads to cardiovascular, cerebrovascular and renal complications. Despite the availability of multitudes of anti-hypertensive drugs, the percentage of patients achieving optimal control of hypertension has remained disappointingly low.

Resistant hypertension (rHT) is defined as the failure to achieve target BP despite concurrent use of antihypertensive drugs of different classes, with one of them being diuretics. The reported prevalence of this condition ranged from 5 to 30%. Lifestyle modification, enhancing drug compliance, treating of secondary causes, or adding mineralocorticoid receptor antagonist such as spironolactone or eplerenone are well established strategies to treat resistant hypertension.

Besides factors such as, activated sympathetic nervous system (SNS) and increased sympathetic outflow was thought to contribute to the development of rHT as well. Autonomic sympathectomy by way of endovascular renal denervation (RDN) was once a hopeful candidate as an adjuvant treatment for patients with rHT and it had shown signals of efficacy in early trials. However, the blood-pressure lowering efficacy was not demonstrated in the larger-scaled, randomized, sham- controlled SYMPLICITY HTN-3 trial. One possible explanation of the lack of efficacy of RDN in this trial was the lower-than-expected BP responses in the RDN group and higher than-expected BP reduction in the control group which raised the speculation that some of the patients recruited were not true rHT as the trial intended to include. The suboptimal anti-hypertensive efficacy of RDN in HTN-3 was also partly attributed to the design of the first-generation RDN catheter, in which only a single electrode is deployed and might not offer sufficient sympathetic denervation as less than half of patients in the SYMPLICITY HTN-3 received 4 quadrants ablation.

The second generation SYMPLICITY RDN catheterTM has 4 times electrodes that are arranged in spirally in 90-degree intervals. Theoretically, the newer generation catheter can provide more efficient and extensive denervation in a shorter period of time. Its efficacy was confirmed in SYMPLICITY HTN ON-MED and OFF-MED trial, which confirmed a consistent and durable BP reduction that lasted into 36 months with or without adjuvant anti-hypertensive drugs.

BP reduction is only one of the effects of RDN. Previous observational studies of the first generation RDN catheter have shown an inconsistent effect of RDN in left ventricular (LV) remodelling, arrythmia modulation, arterial de-stiffening and quality of life. No report of these effects has been published with the newer generation catheter. Furthermore, vigorous efforts have been put into searching for clinical predictors that can identify patients in whom the BP reduction effect of RDN is most significant.

This study aims to investigate the systemic effects of RDN using the new generation SYMLICITY RDN catheterTM in patients with rHT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age >18.
2. Subject (or legal guardian) understands the study procedures and provides written informed consent.
3. Subject is recruited for Transcatheter Renal Denervation Procedure.

Exclusion Criteria:

There is no exclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a feasibility study, small sample size serves as a proof of concept
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
Changes in SBP and DBP as measured by office BP measurement and by 24 hours ABPM | 24 hours
Changes in Echocardiographic parameters including LV wall thickness, LV mass, LV dimension, LV systolic function, LV diastolic function, LV global longitudinal strain, LA volume, LA strain, descending aortic circumferential strain, and RV function. | 24 hours
Changes in arterial stiffness as measured by brachial pulse wave velocity. | 24 hours
Changes in serum renin/aldosterone level and 24 hours urine metanephrines | 24 hours

SECONDARY OUTCOMES:
Change in number and dose of anti-hypertensives | 6-months
Change in renal function as measured by estimated GFR and urine albumin creatine ratio. | 6-months
Change in Patient's SF 36 survey | 6-months
Change in Hba1c | 6-months
MACE including occurrence of new myocardial infarction or stroke. | 6-months
All course morality | 6-months
Change in renal function as measured by urine albumin creatine ratio. | 6-months
Change in LDL and HDL | 6-months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Result] Whitworth JA; World Health Organization, International Society of Hypertension Writing Group. 2003 World Health Organization (WHO)/International Society of Hypertension (ISH) statement on management of hypertension. J Hypertens. 2003 Nov;21(11):1983-92. doi: 10.1097/00004872-200311000-00002. PMID 14597836
- [Result] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Result] Carey RM, Calhoun DA, Bakris GL, Brook RD, Daugherty SL, Dennison-Himmelfarb CR, Egan BM, Flack JM, Gidding SS, Judd E, Lackland DT, Laffer CL, Newton-Cheh C, Smith SM, Taler SJ, Textor SC, Turan TN, White WB; American Heart Association Professional/Public Education and Publications Committee of the Council on Hypertension; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Genomic and Precision Medicine; Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Stroke Council. Resistant Hypertension: Detection, Evaluation, and Management: A Scientific Statement From the American Heart Association. Hypertension. 2018 Nov;72(5):e53-e90. doi: 10.1161/HYP.0000000000000084. PMID 30354828
- [Result] Carey RM, Sakhuja S, Calhoun DA, Whelton PK, Muntner P. Prevalence of Apparent Treatment-Resistant Hypertension in the United States. Hypertension. 2019 Feb;73(2):424-431. doi: 10.1161/HYPERTENSIONAHA.118.12191. PMID 30580690
- [Result] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Result] Anderson EA, Sinkey CA, Lawton WJ, Mark AL. Elevated sympathetic nerve activity in borderline hypertensive humans. Evidence from direct intraneural recordings. Hypertension. 1989 Aug;14(2):177-83. doi: 10.1161/01.hyp.14.2.177. PMID 2759678
- [Result] SMITHWICK RH, THOMPSON JE. Splanchnicectomy for essential hypertension; results in 1,266 cases. J Am Med Assoc. 1953 Aug 15;152(16):1501-4. doi: 10.1001/jama.1953.03690160001001. No abstract available. PMID 13061307
- [Result] Symplicity HTN-1 Investigators. Catheter-based renal sympathetic denervation for resistant hypertension: durability of blood pressure reduction out to 24 months. Hypertension. 2011 May;57(5):911-7. doi: 10.1161/HYPERTENSIONAHA.110.163014. Epub 2011 Mar 14. PMID 21403086
- [Result] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Result] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Result] Tam GM, Yan BP, Shetty SV, Lam YY. Transcatheter renal artery sympathetic denervation for resistant hypertension: an old paradigm revisited. Int J Cardiol. 2013 Apr 15;164(3):277-81. doi: 10.1016/j.ijcard.2012.01.048. Epub 2012 Feb 14. PMID 22336259
- [Result] Bakris GL, Townsend RR, Flack JM, Brar S, Cohen SA, D'Agostino R, Kandzari DE, Katzen BT, Leon MB, Mauri L, Negoita M, O'Neill WW, Oparil S, Rocha-Singh K, Bhatt DL; SYMPLICITY HTN-3 Investigators. 12-month blood pressure results of catheter-based renal artery denervation for resistant hypertension: the SYMPLICITY HTN-3 trial. J Am Coll Cardiol. 2015 Apr 7;65(13):1314-1321. doi: 10.1016/j.jacc.2015.01.037. PMID 25835443
- [Result] Kandzari DE, Bhatt DL, Brar S, Devireddy CM, Esler M, Fahy M, Flack JM, Katzen BT, Lea J, Lee DP, Leon MB, Ma A, Massaro J, Mauri L, Oparil S, O'Neill WW, Patel MR, Rocha-Singh K, Sobotka PA, Svetkey L, Townsend RR, Bakris GL. Predictors of blood pressure response in the SYMPLICITY HTN-3 trial. Eur Heart J. 2015 Jan 21;36(4):219-27. doi: 10.1093/eurheartj/ehu441. Epub 2014 Nov 16. PMID 25400162
- [Result] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Result] Bohm M, Kario K, Kandzari DE, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Konstantinidis D, Choi JW, East C, Lee DP, Ma A, Ewen S, Cohen DL, Wilensky R, Devireddy CM, Lea J, Schmid A, Weil J, Agdirlioglu T, Reedus D, Jefferson BK, Reyes D, D'Souza R, Sharp ASP, Sharif F, Fahy M, DeBruin V, Cohen SA, Brar S, Townsend RR; SPYRAL HTN-OFF MED Pivotal Investigators. Efficacy of catheter-based renal denervation in the absence of antihypertensive medications (SPYRAL HTN-OFF MED Pivotal): a multicentre, randomised, sham-controlled trial. Lancet. 2020 May 2;395(10234):1444-1451. doi: 10.1016/S0140-6736(20)30554-7. Epub 2020 Mar 29. PMID 32234534
- [Result] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Result] Mahfoud F, Kandzari DE, Kario K, Townsend RR, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Dimitriadis K, Choi JW, East C, D'Souza R, Sharp ASP, Ewen S, Walton A, Hopper I, Brar S, McKenna P, Fahy M, Bohm M. Long-term efficacy and safety of renal denervation in the presence of antihypertensive drugs (SPYRAL HTN-ON MED): a randomised, sham-controlled trial. Lancet. 2022 Apr 9;399(10333):1401-1410. doi: 10.1016/S0140-6736(22)00455-X. Epub 2022 Apr 4. PMID 35390320
- [Result] Brandt MC, Mahfoud F, Reda S, Schirmer SH, Erdmann E, Bohm M, Hoppe UC. Renal sympathetic denervation reduces left ventricular hypertrophy and improves cardiac function in patients with resistant hypertension. J Am Coll Cardiol. 2012 Mar 6;59(10):901-9. doi: 10.1016/j.jacc.2011.11.034. PMID 22381425
- [Result] Schirmer SH, Sayed MM, Reil JC, Ukena C, Linz D, Kindermann M, Laufs U, Mahfoud F, Bohm M. Improvements in left ventricular hypertrophy and diastolic function following renal denervation: effects beyond blood pressure and heart rate reduction. J Am Coll Cardiol. 2014 May 13;63(18):1916-23. doi: 10.1016/j.jacc.2013.10.073. Epub 2013 Dec 4. PMID 24315919
- [Result] Mahfoud F, Urban D, Teller D, Linz D, Stawowy P, Hassel JH, Fries P, Dreysse S, Wellnhofer E, Schneider G, Buecker A, Schneeweis C, Doltra A, Schlaich MP, Esler MD, Fleck E, Bohm M, Kelle S. Effect of renal denervation on left ventricular mass and function in patients with resistant hypertension: data from a multi-centre cardiovascular magnetic resonance imaging trial. Eur Heart J. 2014 Sep 1;35(33):2224-31b. doi: 10.1093/eurheartj/ehu093. Epub 2014 Mar 6. PMID 24603307
- [Result] Ukena C, Bauer A, Mahfoud F, Schreieck J, Neuberger HR, Eick C, Sobotka PA, Gawaz M, Bohm M. Renal sympathetic denervation for treatment of electrical storm: first-in-man experience. Clin Res Cardiol. 2012 Jan;101(1):63-7. doi: 10.1007/s00392-011-0365-5. Epub 2011 Sep 29. PMID 21960416
- [Result] Linz D, Mahfoud F, Schotten U, Ukena C, Neuberger HR, Wirth K, Bohm M. Renal sympathetic denervation suppresses postapneic blood pressure rises and atrial fibrillation in a model for sleep apnea. Hypertension. 2012 Jul;60(1):172-8. doi: 10.1161/HYPERTENSIONAHA.112.191965. Epub 2012 May 14. PMID 22585944
- [Result] Peters CD, Mathiassen ON, Vase H, Bech Norgaard J, Christensen KL, Schroeder AP, Rickers HJVH, Opstrup UK, Poulsen PL, Langfeldt S, Andersen G, Hansen KW, Botker HE, Engholm M, Bertelsen JB, Pedersen EB, Kaltoft A, Buus NH. The effect of renal denervation on arterial stiffness, central blood pressure and heart rate variability in treatment resistant essential hypertension: a substudy of a randomized sham-controlled double-blinded trial (the ReSET trial). Blood Press. 2017 Dec;26(6):366-380. doi: 10.1080/08037051.2017.1368368. Epub 2017 Aug 23. PMID 28830251
- [Result] Berukstis A, Navickas R, Neverauskaite-Piliponiene G, Ryliskyte L, Misiura J, Vajauskas D, Misonis N, Laucevicius A. Arterial Destiffening Starts Early after Renal Artery Denervation. Int J Hypertens. 2019 Mar 3;2019:3845690. doi: 10.1155/2019/3845690. eCollection 2019. PMID 30941209
- [Result] Krawczyk-Ozog A, Tokarek T, Moczala K, Siudak Z, Dziewierz A, Mielecki W, Gorecki T, Gerba K, Dudek D. Long-term quality of life and clinical outcomes in patients with resistant hypertension treated with renal denervation. Postepy Kardiol Interwencyjnej. 2016;12(4):329-333. doi: 10.5114/aic.2016.63633. Epub 2016 Nov 17. PMID 27980546
- [Result] Mitchell C, Rahko PS, Blauwet LA, Canaday B, Finstuen JA, Foster MC, Horton K, Ogunyankin KO, Palma RA, Velazquez EJ. Guidelines for Performing a Comprehensive Transthoracic Echocardiographic Examination in Adults: Recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2019 Jan;32(1):1-64. doi: 10.1016/j.echo.2018.06.004. Epub 2018 Oct 1. No abstract available. PMID 30282592